CLINICAL TRIAL: NCT01636375
Title: The Influence of Operative Approach on Muscle Atrophy After Total Hip Arthroplasty: A Comparison of Anterior and Posterior Approaches
Brief Title: Comparison of Muscle Atrophy After Direct Anterior & Posterior Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Jose Rodriguez, MD, MD, Director, Center For Joint Preservation & Reconstruction,NorthShoreLIJ/LenoxHill Hospital, Northwell Health
Other Study IDs: MRI DAA/PA
Record Dates: First submitted 2012-06-29; First posted 2012-07-10 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Direct Anterior Approach
- Posterior Approach

SUMMARY:
This project is designed to use MRI to evaluate pre- and post-arthroplasty hips; the specific aims of this project are three-fold. First, the investigators intend to compare the amount of muscle atrophy and tendon damage that occurs around the hip between two commonly-used operative approaches: the direct-anterior approach and the posterior approach. Second, the investigators aim to provide baseline data on the amount of muscle atrophy and tendon damage that should reasonably be expected to occur with both of these approaches. Third, the investigators will document the degree of recovery of the periprosthetic soft tissues post-surgery in both patient groups.

The investigators first hypothesis is that the posterior approach will demonstrate significantly more damage to the abductors, piriformis, and short external rotators than the direct anterior approach, which will demonstrate minimal soft tissue damage. The investigators second hypothesis is that both surgical approaches will cause some degree of baseline muscle damage and atrophy, in a predictable pattern. The investigators third hypothesis is that each of the surgical approaches inherently cause some degree of soft tissue damage, and that the periprosthetic soft tissues that are incised during the surgical exposure will recover in a predictable pattern which is consistent but unique within each group

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective, primary total hip arthroplasty
2. Use of Cementless Total Hip components
3. Preoperative diagnosis of degenerative joint disease secondary to osteoarthritis

Exclusion Criteria:

1. Prior surgery on the affected hip
2. No implanted medical devices or metallic debris in the patient which will preclude use of MRI
3. patients must be able to participate in standard post-arthroplasty rehabilitation protocols.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Total Hip arthroplasty by one of the two fellowship trained arthroplasty surgeons.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-05; Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in muscle volume at 6 weeks | 6 weeks after surgery
  Muscle volume will be recorded in MRI images with specialized software (external rotators,tensor fascia lata, rectus femoris,gluteus medius and minimus)
Change from baseline in muscle volume at 6 months | 6 months after surgery

SECONDARY OUTCOMES:
Change in Fatty atrophy of muscles from baseline at 6weeks | 6 weeks after surgery
  Qualitative assessment of fatty atrophy
tendon damage | 6 weeks after surgery
  Qualitative assessment of tendon damage on MRI
Change in fatty atrophy of muscles from baseline at 6 months | 6 months after surgery
Tendon damage | 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Rodriguez, MD, Principal Investigator — NorthShoreLIJ/LenoxHill Hospital
Locations (1):
- NorthShoreLIJ/LenoxHill Hospital, New York, New York, United States